CLINICAL TRIAL: NCT07104773
Title: Clinical Investigation of Proclear® 1 Day and MyDay® Sphere Contact Lenses
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision International Limited (CVIL) (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-169
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-06

CONDITIONS: Ametropia; Myopia
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Lens (omafilcon A) (Experimental): All participants will wear Control Lens for 15 minutes (Period 1).
  Interventions: Device: Control Lens (omafilcon A)
- Test Lens (stenfilcon A) (Experimental): All participants will wear Test Lens for 15 minutes (Period 2).
  Interventions: Device: Test Lens (stenfilcon A)

INTERVENTIONS:
Device: Control Lens (omafilcon A) — 15 minutes of daily wear
  Arms: Control Lens (omafilcon A)
Device: Test Lens (stenfilcon A) — 15 minutes of daily wear
  Arms: Test Lens (stenfilcon A)

SUMMARY:
The aim of this study is to evaluate and compare the performance of two soft contact lenses.

DETAILED DESCRIPTION:
The aim of this study is to evaluate and compare the performance of a hydrogel lens and a silicone hydrogel lens in existing soft lens wearers.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 18 years of age and have capacity to consent;
2. Have understood and signed an information consent form;
3. Are an adapted soft contact lens wearer (worn for at least 3 months);
4. Have a contact lens prescription of -1.00DS to -6.00DS (inclusive) in each eye;
5. Have a refraction with a cylinder component of no more than -0.75DC in each eye;
6. Can achieve a best spectacle-corrected visual acuity in each eye of +0.10 logMAR or better.

Exclusion Criteria:

1. Participation in a contact lens or contact lens care product clinical trial in the previous 30 days;
2. Have any known active anterior segment disease and/or infection or slit lamp findings that would contraindicate contact lens wear;
3. Have a systemic condition that would contraindicate contact lens wear;
4. Are using any systemic or topical medications that would contraindicate contact lens wear;
5. Have known sensitivity to the diagnostic fluorescein sodium to be used in the study;
6. Are an employee of the study site (Centre for Ocular Research & Education) and directly involved in the study (ie. on the delegation log).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Subjective Comfort Rating | At the end of 15 minutes of daily wear
  The primary outcome of this study is lens comfort on a scale of 0-100 (0= worst, 100=best).

CONTACTS AND LOCATIONS:
Overall Officials: Jill Woods, MSc, MCOptom, Principal Investigator — Centre of Ocular Research and Education
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada